CLINICAL TRIAL: NCT06351072
Title: Correlation Between qNOX Values of the CONOX Monitor and Analgesia Nociception Index (ANI) Values During General Anesthesia Conducted With Propofol and Remifentanil TCI
Brief Title: Correlation Between qNOX and Analgesia Nociception Index (ANI) Values During General Anesthesia
Acronym: ANI
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Federico Linassi, MD, principal invesigator, University of Padova
Other Study IDs: NOXANI
Record Dates: First submitted 2024-03-25; First posted 2024-04-08 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
qNOX and ANI are two indexes evaluting the analgesia conduction during general anesthesia.

No trials have compared them, so with this trial authors want to explore the correlations between them.

DETAILED DESCRIPTION:
qNOX and ANI are two indexes evaluting the anaglesia conduction during general anesthesia.

Even if the aim is the same (to measure the nociception level) these indexes utilize different algorithm: the qNOX is derived by the electroencephalogrm (EEG), the ANI is derived by heart rate variation.

No trials have compared them, so with this trial authors want to explore the correlations between them, and if altered values of one of them is stronger related to postoperative pain and delirium.

ELIGIBILITY:
Inclusion Criteria:

* Undergo general anaesthesia with Targeted Controlled Infusion of Propofol (Eleveld model) and remifentanil (Eleveld model)

Exclusion Criteria:

* Neurological disease
* Psychiatric disease
* Obesity
* Regional anesthesia performed

Ages: 18 Years to 90 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women undergoing brast cancer surgery with general anesthesia with Propofol and remifentanil TCI will be recruited
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Correlation between qNOX and ANI values | qNOX, ANI, pupoillometry values, propofol and remifentanil concentration during induction, intubation, after post-tetanic count at the trend-of-four and maintenance phase of general anesthesia detected with target controlled inusion will be paired.
  qNOX and ANI values will be compared to check the correspondance in evaluting analgesia level

SECONDARY OUTCOMES:
Correlation between qNOX from CONOX and Analgesia nocicpetion index (ANI) values and postoperative pain | qNOX, ANI and remifentanil concentrations recorded during induction, intubation and maintenance phase of general anesthesia will be related to postoperative pain, evalued with NRS score after 24 hours
  Evaluate if qNOX or ANI values relate to postoperative pain
Correlation between qNOX from CONOX and analgesia nocicpetion index (ANI) values and postoperative delirium | qNOX, ANI and remifentanil concentrations recorded during induction, intubation and maintenance phase of general anesthesia will be related to postoperative delirium, evaluated with CAM and 4AT score after 24 hours
  Evaluate if qNOX or ANI values relate to postoperative delirium

CONTACTS AND LOCATIONS:
Locations (1):
- Treviso Regional Hospital, Treviso, TV, Italy

IPD SHARING:
Plan to Share IPD: Undecided